CLINICAL TRIAL: NCT06346691
Title: Bronchodilator Effect of Oral Doxofylline and Procaterol in Chronic Obstructive Pulmonary Disease : a Randomized Crossover Study
Brief Title: Effects of Oral Doxofylline and Procaterol on Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Narongkorn Saiphoklang, MD, Associate Professor, Thammasat University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MTU-EC-IM-0-235/66
Record Dates: First submitted 2024-03-28; First posted 2024-04-04 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: COPD
Keywords: Chronic obstructive pulmonary disease; COPD; Bronchodilator; Doxofylline; Procaterol; Pulmonary function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — doxofylline; Procaterol

STUDY DESIGN:
Intervention Model Description: Crossover randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doxofylline arm (Experimental): Doxofylline 400 mg oral twice daily for 4 weeks
  Interventions: Drug: Doxofylline
- Procaterol arm (Active Comparator): Procaterol 50 mcg oral twice daily for 4 weeks
  Interventions: Drug: Procaterol

INTERVENTIONS:
Drug: Doxofylline — Each patient received 4 weeks of treatment with either doxofylline or procaterol followed by a 2-week washout period, and then 4 weeks of treatment with the other drug.
  Arms: Doxofylline arm
Drug: Procaterol — Each patient received 4 weeks of treatment with either doxofylline or procaterol followed by a 2-week washout period, and then 4 weeks of treatment with the other drug.
  Arms: Procaterol arm

SUMMARY:
The goal of this clinical trial is to determine if doxofylline and procaterol are effective in treating patients with stable chronic obstructive pulmonary disease (COPD). It will also assess the safety of both drugs.

The main questions it aims to answer are:

* Does doxofylline demonstrate a comparable bronchodilator effect to procaterol in COPD participants?
* What medical problems do participants experience when taking doxofylline and procaterol?"

DETAILED DESCRIPTION:
This study is a randomized crossover study. COPD patients aged 40 years or older with stable disease were included. Each patient received 4 weeks of treatment with either doxofylline or procaterol followed by a 2-week washout period, and then 4 weeks of treatment with the other drug. Respiratory symptoms were assessed by modified Medical Research Council (mMRC) dyspnea scale and COPD Assessment Test (CAT). Pulmonary functions were assessed by spirometry with bronchodilator testing, and adverse events were recorded. Spirometry data including forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), and forced expiratory flow at 25-75% of FVC (FEF25-75) were also collected.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis confirmed by spirometry (post-bronchodilator FEV1/FVC < 70%)
* Aged 40 years or older
* Smoking 10 pack-years or more
* Postbronchodilator FEV1 < 80%

Exclusion Criteria:

* History of COPD exacerbation within 3 months
* Oral or intravenous corticosteroid treatment within 6 weeks
* Oral bronchodilators e.g. doxofylline, theophylline, procaterol, or salbutamol within 1 week before randomization
* Asthma
* Tracheostomy, invasive or noninvasive mechanical ventilation
* Inability to perform spirometry or 6-minute walk test
* Pregnant or breastfeeding women

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) | At the day of randomization (week 0), week 4, week 6, and week 8 of the study
  Postbronchodilator FEV1
Forced vital capacity (FVC) | At the day of randomization (week 0), week 4, week 6, and week 8 of the study
  Postbronchodilator FVC
Forced expiratory flow at 25-75% of FVC (FEF25-75) | At the day of randomization (week 0), week 4, week 6, and week 8 of the study
  Postbronchodilator FEF25-75

SECONDARY OUTCOMES:
modified Medical Research Council (mMRC) score | At the day of randomization (week 0), week 4, week 6, and week 8 of the study
  Scores range from 0 to 4, with higher scores indicating a worse outcome
COPD Assessment Test (CAT) | At the day of randomization (week 0), week 4, week 6, and week 8 of the study
  Scores range from 0 to 40, with higher scores indicating a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Narongkorn Saiphoklang, MD, Principal Investigator — Thammasat University Faculty of Medicine
Locations (1):
- Narongkorn Saiphoklang, Klongluang, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) and documents will be available for sharing immediately after publication for a period of 2 years.
Supporting Information: Study Protocol, SAP, CSR